CLINICAL TRIAL: NCT02571361
Title: PAracetamol and NSAID in Combination: A Randomised, Blinded, Parallel, 4-group Clinical Trial
Acronym: PANSAID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Hägi-Pedersen (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor-Investigator, Daniel Hägi-Pedersen, Consultant, Naestved Hospital
Organization: Naestved Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM2-KHT-2015 - v2; 2015-002239-16 (EudraCT Number)
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Pain, Postoperative
Keywords: Acetaminophen; Ibuprofen; Arthroplasty, Replacement, Hip
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A: (Active Comparator): Paracetamol 1g + ibuprofen 400 mg orally starting 1 hour before surgery and given with 6-hour intervals (+/- 1 hour) i.e. a total of 4 times the first 24 hours postoperative.
  Interventions: Drug: Paracetamol (1g x 4); Drug: Ibuprofen (400 mg x 4)
- Treatment B: (Active Comparator): Paracetamol 1g + placebo orally starting 1 hour before surgery and given with 6-hour intervals (+/- 1 hour) i.e. a total of 4 times the first 24 hours postoperative.
  Interventions: Drug: Paracetamol (1g x 4); Drug: Placebo (x4)
- Treatment C: (Active Comparator): Placebo + ibuprofen 400 mg orally starting 1 hour before surgery and given with 6-hour intervals (+/- 1 hour) i.e. a total of 4 times the first 24 hours postoperative.
  Interventions: Drug: Ibuprofen (400 mg x 4); Drug: Placebo (x4)
- Treatment D: (Active Comparator): Paracetamol 0,5 g + ibuprofen 200 mg orally starting 1 hour before surgery and given with 6-hour intervals (+/- 1 hour) i.e. a total of 4 times the first 24 hours postoperative.
  Interventions: Drug: Paracetamol (0,5 g x 4); Drug: Ibuprofen (200 mg x 4)

INTERVENTIONS:
Drug: Paracetamol (1g x 4) — Dose of 1 g given in 6 hour intervals the first 24 hours postoperatively
  Other Names: Acetaminophen
  Arms: Treatment A:; Treatment B:
Drug: Ibuprofen (400 mg x 4) — Dose of 400 mg given in 6 hour intervals the first 24 hours postoperatively
  Arms: Treatment A:; Treatment C:
Drug: Paracetamol (0,5 g x 4) — Dose of 0,5 g given in 6 hour intervals the first 24 hours postoperatively
  Other Names: Acetaminophen
  Arms: Treatment D:
Drug: Ibuprofen (200 mg x 4) — Dose of 200 mg given in 6 hour intervals the first 24 hours postoperatively
  Arms: Treatment D:
Drug: Placebo (x4) — Given in 6 hour intervals the first 24 hours postoperatively
  Arms: Treatment B:; Treatment C:

SUMMARY:
Trial name: PAracetamol and NSAID in combination: A randomised, blinded, parallel, 4-group clinical trial

Trial acronym: PANSAID

Background: Effective postoperative pain management is essential for the well-being and rehabilitation of the surgical patient. No "gold standard" exists after total hip arthroplasty (THA) and combinations of different non-opioid medications are used with virtually no evidence for additional analgesic efficacy compared to monotherapy.

Objectives: The objective of this trial is to investigate the analgesic effects and safety of paracetamol and ibuprofen and their combination in different dosages after THA.

Intervention: Patients are randomised to 4 groups: A) paracetamol 1 g x 4 and ibuprofen 400 mg x 4; B) paracetamol 1 g x 4 and placebo (ibuprofen); C) placebo (paracetamol) and ibuprofen 400 mg x 4; and D) paracetamol 0,5 g x 4 and ibuprofen 200 mg.

Design: Placebo controlled, parallel 4-group, multicentre trial with adequate centralised computer-generated allocation sequence and allocation concealment with varying block size and stratification by site. Blinding of assessor, investigator, caregivers, patients, and statisticians.

Sample size: 556 eligible patients are needed to detect a difference of 10 mg morphine the first postoperative day with a standard deviation of 20 mg and a type 1 error rate of 0,004 (two-sided) and a type 2 error rate of 0,10.

DETAILED DESCRIPTION:
Trial name: PAracetamol and NSAID in combination: A randomised, blinded, parallel, 4-group clinical trial

Trial acronym: PANSAID

Background: Effective postoperative pain management is essential for the well-being and rehabilitation of the surgical patient. No "gold standard" exists after total hip arthroplasty (THA) and combinations of different non-opioid medications are used with virtually no evidence for additional analgesic efficacy compared to monotherapy.

Objectives: The objective of this trial is to investigate the analgesic effects and safety of paracetamol and ibuprofen and their combination in different dosages after THA.

Intervention: Patients are randomised to 4 groups: A) paracetamol 1 g x 4 and ibuprofen 400 mg x 4; B) paracetamol 1 g x 4 and placebo (ibuprofen); C) placebo (paracetamol) and ibuprofen 400 mg x 4; and D) paracetamol 0,5 g x 4 and ibuprofen 200 mg.

Design: Placebo controlled, parallel 4-group, multicentre trial with adequate centralised computer-generated allocation sequence and allocation concealment with varying block size and stratification by site. Blinding of assessor, investigator, caregivers, patients, and statisticians.

Sample size: 556 eligible patients are needed to detect a difference of 10 mg morphine the first postoperative day with a standard deviation of 20 mg and a type 1 error rate of 0,004 (two-sided) and a type 2 error rate of 0,10.

Sub-studies: We preplan the following sub-studies. :

1. A subgroup analysis of benefit outcomes (pain and opioid consumption) with respect to the following sub-groups: sex, age (below vs above 65 years old), ASA-score (I+II vs III), Use of analgesic medication before surgery (none vs any) and anaesthetic technique (general anaesthesia vs. spinal anaesthesia). Please find a detailed protocol at www.pansaid.dk
2. A subgroup analysis of harm (serious adverse events and adverse events) with respect to the following groups sex, age (below vs above 65 years old), use of NSAIDs before surgery, and ASA-score (I+II vs III). Please find a detailed protocol at www.pansaid.dk
3. Longer follow-up than the specified 90 days (1 year)
4. An analysis of the association between VAS-scores and opioid consumption
5. Time-to-event analyses regarding use of PCA-morphine
6. An analysis of the association between preoperative analgesic use and pain/morphine consumption
7. An analysis of the individual patients: how many will achieve "no worse than mild pain" (NRS<3). Please find a detailed protocol at www.pansaid.dk

More sub-studies may be performed post-hoc and they will be clearly identified as such.

Oversight of amendments and approvals Protocol version 2: Approved 12 August 2015: First approved version of the trial protocol

Protocol version 3: Approved 21 January 2016: Clarification of what happens in case of an SAE and definition of major protocol violations

Protocol version 4: Approved 15 June 2016: Clarification of the primary outcome, clarification that steroids are not permitted in the intervention period, and addition of an exploratory outcome (dizziness)

Protocol version 5: Approved 21 December 2016: Clarification of the exclusion criteria of contraindication to paracetamol and addition of stub-studies

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral, primary Total Hip Arthroplasty (THA)
* Age > 18
* ASA 1-3.
* BMI > 18 and < 40
* Women in the fertile age must have negative urine HCG pregnancy test
* Patients who gave their written informed consent to participating in the trial after having fully understood the contents of the protocol and restrictions.

Exclusion Criteria:

* Patients who cannot cooperate with the trial.
* Concomitant participation in another trial
* Patients who cannot understand or speak Danish.
* Daily use of strong opioids (tramadol and codein are accepted)
* Patients with allergy to the medicines used in the trial.
* Contraindications against NSAID, for example previous ulcer, heart failure, liver failure, or renal failure (eGRF < 60 ml/kg/1,73m2), known thrombocytopenia (<100 mia/L)
* Patients suffering from alcohol and/or drug abuse - based on the investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2015-11; Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption the first 24 hours postoperatively | 0-24 hours postoperatively
  Total need for morphine administered as BOTH patient controlled analgesia (PCA) for the first 24 hours postoperatively AND supplemental morphine administered at the post-anaesthesia unit the first hour postoperatively. Bolus 2.0 mg; lockout: 10 min
Serious adverse events | 0-90 days postoperatively
  Serious adverse events, including death, within 90 days after surgery defined as SAE (according to ICH-GCP-guidelines) except "prolongation of hospitalisation"

SECONDARY OUTCOMES:
Pain during movement at 6 hours postoperatively (visual analogue scale) | 6 hours postoperatively
  Pain scores (visual analogue scale (VAS)) with active 30 degrees flexion of the hip at 6 hours postoperatively. No pain = 0; worst imaginable pain = 100
Pain during movement at 24 hours postoperatively (visual analogue scale) | 24 hours postoperatively
  Pain scores (visual analogue scale (VAS)) with active 30 degrees flexion of the hip at 24 hours postoperatively. No pain = 0; worst imaginable pain = 100
Pain at rest at 6 hours postoperatively (visual analogue scale) | 6 hours postoperatively
  Pain scores (visual analogue scale (VAS)) at rest at 6 hours postoperatively. No pain = 0; worst imaginable pain = 100
Pain at rest at 24 hours postoperatively (visual analogue scale) | 24 hours postoperatively
  Pain scores (visual analogue scale (VAS)) at rest at 24 hours postoperatively. No pain = 0; worst imaginable pain = 100
Adverse events | 0-24 hours postoperatively
  Number of patients with one or more adverse events in the intervention period (0-24 hours)

OTHER OUTCOMES:
Nausea at 6 hours postoperatively (Verbal rating scale) | 6 hours postoperatively
  Level of nausea at 6 hours postoperatively. Verbal rating scale: none, mild, moderate or severe
Nausea at 24 hours postoperatively (Verbal rating scale) | 24 hours postoperatively
  Level of nausea at 24 hours postoperatively. Verbal rating scale: none, mild, moderate or severe
Vomiting the first 24 hours postoperatively | 0-24 hours postoperatively
  Number of vomiting episodes (0-24 hours) measured in the periods 0-6 and 6-24 hours postoperatively
Anti-emetic treatment the first 24 hours postoperatively | 0-24 hours postoperatively
  Consumption of ondansetron in the period 0-24 hours postoperatively
Sedation at 6 hours postoperatively (Verbal rating scale) | 6 hours postoperatively
  Level of sedation at 6 hours postoperatively. Verbal rating scale: none, mild, moderate or severe
Sedation at 24 hours postoperatively (Verbal rating scale) | 24 hours postoperatively
  Level of sedation at 24 hours postoperatively. Verbal rating scale: none, mild, moderate or severe
Blood loss intraoperatively | intraoperatively
  Blood loss during the surgical procedure (intraoperatively)
Days alive and outside hospital within 90 days after surgery. | 0-90 days postoperatively
  Days alive and outside hospital within 90 days after surgery.
Dizziness at 6 hours postoperatively (Verbal rating scale) | 6 hours postoperatively
  Level of dizziness at 6 hours postoperatively. Verbal rating scale: none, mild, moderate or severe
Dizziness at 24 hours postoperatively (Verbal rating scale) | 24 hours postoperatively
  Level of dizziness at 24 hours postoperatively. Verbal rating scale: none, mild, moderate or severe

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hägi-Pedersen, MD, PhD, Study Chair — Department of Anaesthesiology, Næstved Hospital; Kasper H Thybo, MD, Principal Investigator — Department of Anaesthesiology, Næstved Hospital; Ole Mathiesen, MD, PhD, Study Chair — Department of Anaesthesiology, Køge Hospital; Jørgen B Dahl, MD, DMSc, Study Chair — Department of Anaesthesiology, Bispebjerg Hospital; Jørn Wetterslev, MD, PhD, Study Chair — Copenhagen Trial Unit, Center for Clinical Intervention Research; Martin Pohlman, MD, Study Chair — Department of Anaesthesiology, Nykøbing Falster Hospital; Hans Henrik Bülow, MD, Study Chair — Department of Anaesthesiology, Holbæk Hospital
Locations (6):
- Denmark (6):
  - Gildhøj Privathospital, Copenhagen, Brøndby
  - Holbæk Hospital, Holbæk
  - Køge Hospital, Køge
  - Nykøbing Falster Hospital, Nykøbing Falster
  - Næstved Hospital, Næstved
  - Odense University Hospital (OUH), Odense

REFERENCES:
- [Background] Thybo KH, Hagi-Pedersen D, Wetterslev J, Dahl JB, Schroder HM, Bulow HH, Bjorck JG, Mathiesen O. PANSAID - PAracetamol and NSAID in combination: study protocol for a randomised trial. Trials. 2017 Jan 10;18(1):11. doi: 10.1186/s13063-016-1749-7. PMID 28069072
- [Derived] Thybo KH, Hagi-Pedersen D, Dahl JB, Wetterslev J, Nersesjan M, Jakobsen JC, Pedersen NA, Overgaard S, Schroder HM, Schmidt H, Bjorck JG, Skovmand K, Frederiksen R, Buus-Nielsen M, Sorensen CV, Kruuse LS, Lindholm P, Mathiesen O. Effect of Combination of Paracetamol (Acetaminophen) and Ibuprofen vs Either Alone on Patient-Controlled Morphine Consumption in the First 24 Hours After Total Hip Arthroplasty: The PANSAID Randomized Clinical Trial. JAMA. 2019 Feb 12;321(6):562-571. doi: 10.1001/jama.2018.22039. PMID 30747964
- [Derived] Thybo KH, Jakobsen JC, Hagi-Pedersen D, Pedersen NA, Dahl JB, Schroder HM, Bulow HH, Bjorck JG, Overgaard S, Mathiesen O, Wetterslev J. PANSAID-PAracetamol and NSAID in combination: detailed statistical analysis plan for a randomised, blinded, parallel, four-group multicentre clinical trial. Trials. 2017 Oct 10;18(1):465. doi: 10.1186/s13063-017-2203-1. PMID 29017585
- See also: Trial Website — http://www.pansaid.dk